CLINICAL TRIAL: NCT00418132
Title: T Cell Immunity in Collagen Biosynthesis of Scleroderma
Brief Title: Thalidomide for Decreasing Collagen Biosynthesis in People With Progressive Systemic Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early due to difficulties in subject recruitment
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Stephen J. Oliver, MD, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23AR002187 (NIH); K23AR002187 (NIH)
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Scleroderma, Systemic
Keywords: SSc; Systemic Sclerosis; Progressive Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive thalidomide.
  Interventions: Drug: Thalidomide
- 2 (Placebo Comparator): Participants will receive placebo thalidomide.
  Interventions: Drug: Placebo thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide at a dose of 50 mg/day. The dose will be increased to 100 mg/day at Week 2, then to 200 mg/day at Week 4, and finally to 300 mg/day at Week 6.
  Arms: 1
Drug: Placebo thalidomide — Participants will receive placebo thalidomide. The placebo dose will be increased through to Week 6.
  Arms: 2

SUMMARY:
Progressive systemic sclerosis (SSc) is an immune-based disease that causes abnormal connective tissue growth of the skin and internal organs. At this point, there are no effective therapies for treating SSc. Thalidomide is a medication that has been shown to stimulate an immune response that reduces the body's synthesis of collagen, the main component of connective tissue. This study will determine the effectiveness of thalidomide in treating adults with SSc.

DETAILED DESCRIPTION:
Progressive systemic sclerosis (SSc), also known as scleroderma, is a disease of the body's connective tissue. It is characterized by fibrosis of the skin, or formation of scar-like tissue, resulting in progressively increased restriction of joint range of motion. Fibrosis of internal organs also occurs, leading to irregular heart rhythms, acid reflux, and respiratory problems. Unfortunately, no therapies have been developed to effectively treat SSc.

The disease is believed to be an immunological disorder that affects T-helper type 2 (Th2) cells, which stimulate the production of antibodies and interleukin-4 (IL-4), a protein with profibrotic properties. T-helper type 1 (Th1) cells produce interferon-γ (IFN-γ), a protein that prevents fibroblast production of collagen, a primary component of the body's connective tissue. It is possible that shifting the disease's target from the Th2 cells to the Th1 cells may decrease collagen production, and thereby reduce fibrosis. Thalidomide is an immune modulatory drug that has been shown to stimulate production of Th1 cells. This study will evaluate the effectiveness of thalidomide in treating adults with SSc.

Following screening procedures, participants in this 48-week, double-blind study will be randomly assigned to receive placebo or thalidomide at a dose of 50 mg/day. The thalidomide dose will be increased to 100 mg/day at Week 2, then to 200 mg/day at Week 4, and finally to 300 mg/day at Week 6. Participants who experience dose intolerance will immediately switch to the previously tolerated dose. Inpatient hospital visits lasting 2 days will occur at the beginning of the study before starting thalidomide treatment and at Weeks 16 and 48. Assessments and procedures at these visits will include blood and urine collection, a physical exam, a chest X-ray, an electrocardiogram, a skin biopsy, and various questionnaires. Outpatient study visits will occur at Weeks 2, 4, 6, 8, 12, 18, 20 and then every 4 weeks until Week 44. Assessments will include measures of immune function, clinical disease, hypothalamic-pituitary-adrenal axis, and safety. Following the Week 48 inpatient visit, thalidomide will be tapered off over a 2-week period for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of scleroderma
* Agrees to use an effective form of contraception for 1 month prior to study entry, throughout the study, and for 60 days after completing the study
* Positive serum anti-nuclear antibody titer

Exclusion Criteria:

* Systemic sclerosis-like illnesses associated with environmental, ingested, or injected agents or with other connective tissue diseases
* Significant existing damage to any of the following internal organs:

  * Kidneys, defined as a serum creatinine level greater than 2 mg/dl or renal crisis
  * Lungs, defined as needing supplemental oxygen
  * Heart, defined as left ventricular ejection fraction less than or equal to 40%
  * Gut, defined as pseudo-obstruction or malabsorption requiring total parental nutrition
* Concurrent interventional therapy that might independently influence the outcome of this trial (e.g., D-penicillamine, cyclosporine, interferon-γ, methotrexate, or photophorosis)
* Clinically significant and inadequately medically treated concurrent endocrine, blood, liver, lung, or kidney diseases
* Pregnant
* Recent drug or alcohol abuse
* Documented noncompliance
* Significant psychiatric history
* Therapy with another investigational drug within 4 weeks prior to study entry
* Screening laboratory results exceeding the following limits: hemoglobin level less than 7 gm/dl; white blood cell level less than 3,000/nl; platelet count less than 50/nl; alanine aminotransferase (ALT) level greater than 65 U/L; creatinine level greater than 2 mg/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-08; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Collagen mRNA levels in the skin | Measured at Weeks 16 and 48
In vivo collagen production | Measured at Weeks 16 and 48

SECONDARY OUTCOMES:
Immune function | Measured at Weeks 4, 16, and 48
Clinical disease measures | Measured at Weeks 16 and 48
Hypothalamic-Pituitary-Adrenal (HPA) axis measures | Measured at Weeks 16 and 48
Safety measures | Measured at Weeks 4, 16, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Oliver, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine General Clinical Research Center, Bellevue Hospital, New York, New York, United States